CLINICAL TRIAL: NCT07285746
Title: Atelocollagen ＆ Hyaluronic Acid Correlation With Enhancement of Rotator Cuff Healing: Synergistic Effect? 2-Year Results of a Randomized Controlled Trial
Brief Title: Atelocollagen ＆ Hyaluronic Acid Correlation With Enhancement of Rotator Cuff Healing: Synergistic Effect?
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Dongtan Sacred Heart Hospital (Other)
Collaborators: Ministry of Science and ICT, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, JEUNGYEOL JEONG, Associate Professor of Orthopaedics, Hallym University Dongtan Sacred Heart Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HDT 2020-12-003
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff tear; Healing; Atelo collagen; Hyaluronic acid
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Atelo collagen + HA Group (Experimental): Patients receive injections of atelo collagen and HA during arthroscopic rotator cuff repair
  Interventions: Procedure: Atelo collagen injection; Procedure: Hyaluronic acid injection
- HA only Group (Experimental): Patients receive injection of HA during arthroscopic rotator cuff repair
  Interventions: Procedure: Hyaluronic acid injection
- Atelo collagen only Group (Experimental): Patients receive injection of Atelo collagen during arthroscopic rotator cuff repair
  Interventions: Procedure: Atelo collagen injection
- No injection Group (No Intervention): Patients do not receive any injections during arthroscopic rotator cuff repair.

INTERVENTIONS:
Procedure: Atelo collagen injection — Patients receive atelocollagen injection during arthroscopic rotator cuff repair.
  Arms: Atelo collagen + HA Group; Atelo collagen only Group
Procedure: Hyaluronic acid injection — Patients receive hyaluronic acid injection during arthroscopic rotator cuff repair.
  Arms: Atelo collagen + HA Group; HA only Group

SUMMARY:
The purpose of this study is to analyze the correlation between the synergistic effects of atelocollagen and hyaluronic acid (HA) in enhancing rotator cuff healing postoperatively in patients undergoing rotator cuff repair surgery.The main questions it aims to answer are:

* Does atelo Collagen aid in the rotator cuff repair healing process?
* Does hyaluronic acid (HA) aid in the rotator cuff repair healing process?
* Does the combined use of atelo collagen and HA in the rotator cuff repair healing process have a synergistic effect?

The researchers will compare the use of atelo collagen and HA alone with no treatment to determine their effectiveness in rotator cuff healing.

Participants will:

* receive injections of atelo collagen or HA, either alone or in combination, during arthroscopic rotator cuff repair.
* visit the clinic for medical checkups and tests every 3 months, 6 months, 1 year, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75 years
* Scheduled for arthroscopic surgery after an MRI confirmed a diagnosis of rotator cuff tear
* Willing to participate and provide informed consent

Exclusion Criteria:

* Previous surgery on the affected shoulder
* Severe glenohumeral arthritis (Hamada grade ≥ 3)
* Neurological disorder affecting shoulder function
* Massive rotator cuff tear (Tear size ≥ 5 cm)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rotator cuff healing status | 6 and 24 months after surgery
  Assessed by MRI according to Sugaya classification & cuff muscle atrophy ratio

SECONDARY OUTCOMES:
Pain Level | 3 months, 6 months, 12 months and 2 years after surgery
  Measured by Visual Analog Scale (0-10, higher score indicates worse result)
Functional Improvement of the Shoulder | 3 months, 6 months, 12 months, and 2 years after surgery
  Measured by American Shoulder and Elbow Surgeons Score (0-100, higher score indicates better function)
Range of Motion | 3 months, 6 months, 12 months, and 2 years after surgery
  Measured using goniometer for forward elevation and external rotation

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Weeks KD 3rd, Dines JS, Rodeo SA, Bedi A. The basic science behind biologic augmentation of tendon-bone healing: a scientific review. Instr Course Lect. 2014;63:443-50. PMID 24720329
- [Background] Cunningham G, Ladermann A, Denard PJ, Kherad O, Burkhart SS. Correlation Between American Shoulder and Elbow Surgeons and Single Assessment Numerical Evaluation Score After Rotator Cuff or SLAP Repair. Arthroscopy. 2015 Sep;31(9):1688-92. doi: 10.1016/j.arthro.2015.03.010. Epub 2015 Apr 22. PMID 25911388
- [Background] Walsh MR, Nelson BJ, Braman JP, Yonke B, Obermeier M, Raja A, Reams M. Platelet-rich plasma in fibrin matrix to augment rotator cuff repair: a prospective, single-blinded, randomized study with 2-year follow-up. J Shoulder Elbow Surg. 2018 Sep;27(9):1553-1563. doi: 10.1016/j.jse.2018.05.003. Epub 2018 Jul 9. PMID 29996980
- [Result] Kim JH, Kim DJ, Lee HJ, Kim BK, Kim YS. Atelocollagen Injection Improves Tendon Integrity in Partial-Thickness Rotator Cuff Tears: A Prospective Comparative Study. Orthop J Sports Med. 2020 Feb 21;8(2):2325967120904012. doi: 10.1177/2325967120904012. eCollection 2020 Feb. PMID 32128319
- [Result] Honda H, Gotoh M, Kanazawa T, Ohzono H, Nakamura H, Ohta K, Nakamura KI, Fukuda K, Teramura T, Hashimoto T, Shichijo S, Shiba N. Hyaluronic Acid Accelerates Tendon-to-Bone Healing After Rotator Cuff Repair. Am J Sports Med. 2017 Dec;45(14):3322-3330. doi: 10.1177/0363546517720199. Epub 2017 Sep 5. PMID 28872895
- [Result] Suh DS, Lee JK, Yoo JC, Woo SH, Kim GR, Kim JW, Choi NY, Kim Y, Song HS. Atelocollagen Enhances the Healing of Rotator Cuff Tendon in Rabbit Model. Am J Sports Med. 2017 Jul;45(9):2019-2027. doi: 10.1177/0363546517703336. Epub 2017 Jun 6. PMID 28586622
- [Result] Li H, Chen Y, Chen S. Enhancement of rotator cuff tendon-bone healing using bone marrow-stimulating technique along with hyaluronic acid. J Orthop Translat. 2019 Jan 28;17:96-102. doi: 10.1016/j.jot.2019.01.001. eCollection 2019 Apr. PMID 31194057

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT07285746/Prot_SAP_ICF_000.pdf